CLINICAL TRIAL: NCT06089018
Title: Observational Study of Digital Biomarkers of Myotonia and Gait in Adults and Children With Myotonic Dystrophy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Stanford University (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, Tina Duong, Director of Clinical Outcomes Research and Development, Stanford University
Other Study IDs: 62522
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Myotonic Dystrophy 1
Keywords: Myotonic Dystrophy 1; DM1; Digital Biomarkers; Hand Myotonia; Gait; Observational Study; Actigraph; Syde
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Myotonic Dystrophy Type 1: This group will consist of participants with a confirmed genetic diagnosis of DM1 or DM2.
- Healthy Controls: This group will consist of participants without a confirmed genetic diagnosis of DM1 or DM2.

SUMMARY:
The goal of this observational study is to assess movement in individuals with Myotonic Dystrophy Type 1 (DM1) and Type 2 (DM2) using digital biomarker tools. The long-term aim of this study is to incorporate these outcomes into clinical trials of DM1 and DM2 therapies. Participants will complete a series of assessments that allow for researchers to measure hand myotonia and walking quality, including a Video Hand Opening Test (VHOT), grip strength, 10 meter walk/run test, 6 minute walk test, Timed Up and Go (TUG), Motor Function Measures-32 (MFM-32) test, and more. These assessments may be recorded to detect and map participants motion and walking patterns. Several patient reported outcome (PROs) questionnaires will also be recorded. Participants may also be asked to monitor exercise and sleep activity at home using an Actigraph wearable device. This study is divided into 2 parts: Part A consists of a single visit. Part B consists of a 1-year longitudinal study with 3 clinical follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Age 12-90 years old at the time of informed consent
* Genetic confirmation of DM1 or DM2
* Ability to comply with study assessments
* Clinically apparent myotonia equivalent to hand opening time of at least 2 seconds, in the opinion of the Investigator
* Ambulatory (orthoses allowed, canes and walkers not allowed) and able to walk at least 25 meters at screening

Exclusion Criteria:

* Ongoing medical condition (e.g. wasting or cachexia, severe anemia) that would, in the opinion of the Investigator, interfere with the conduct or assessments of the study
* Significant cognitive impairment, clinical dementia, or unstable psychiatric illness, including psychosis, suicidal ideation, suicide attempt, or untreated major depression ≤ 90 days of screening, which in the opinion of the Investigator may interfere with the study procedures
* Treatment with an investigational drug, biologic agent, or device within one month of screening, or 5 half-lives of investigational agent, whichever is longer
* Inability to comply with study requirements
* Other unspecified reasons that, in the opinion of the Investigator or the Sponsor, make the participant unsuitable for enrolment

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with genetic confirmation of DM1 or DM2, or with DMPK CTG repeat length >100, or CCTG repeat length >100. We will recruit from our database of subjects with Myotonic Dystrophy that have been seen in the Stanford clinic in the past 5 years. Other neuromuscular specialists in the Bay Area will be informed and will be asked to refer patients to us for the study. We work closely with the Myotonic Dystrophy Foundation, Muscular Dystrophy Foundation, and Myotonic Dystrophy support groups and will spread the word about the study through these as well. We have a separate database of healthy controls that have expressed interest in our research. We will enroll healthy controls via this database, or from laboratory personnel who volunteer.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2022-09-10 (Actual); Primary Completion 2024-09-10 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
Video Hand Opening Time (VHOT) | Baseline through month 12
  With the use of wearable devices, the participant will be asked to open their hand from a fully fisted position as quickly as possible. This assessment will be recorded with a camera as well.
Grip Strength | Baseline through month 12
  Requires a participant to squeeze a device as hard as possible, while the research team measures how much force is produced.
Motor Function Measures (MFM-32) | Baseline through month 12
  This is a motor function test to assess how well a participant can walk, move, and use their hands. The test includes tasks such as reaching and picking up objects, putting out hands, and taking a step.
10 Meter Walk/Run Test | Baseline through month 12
  From a standing start, the participant is asked to go 10 meters as quickly as possible, either by walking or running. Ankle braces and orthotics may be used.
6 Minute Walk Test | Baseline through month 12
  Participant is asked to walk as far as possible within 6 minutes. The participant will be instructed to walk at their normal pace towards a cone, then turn around, continuing to do so for 6 minutes, Ankle braces and orthoses may be used.
Timed Up and Go (TUG) | Baseline through month 12
  The participant will be asked to rise from a chair, walk 3 meters, turn around, return to the chair and sit down. The test will be performed twice, once at a comfortable pace and once at a maximal pace. Assistive devices, orthoses and ankle braces may be used.
Time to Ascend and Descend 4 Stairs | Baseline through month 12
  In this task, the participant will climb up and down 4 stairs as quickly as possible. The manner of ascent/descent and the use of railings will be assessed using quality grades.
Timed Supine to Sit | Baseline through month 12
  This functional assessment is used to assess axial strength. The participant will be asked to move from supine position to sitting on the edge of a table as quickly as possible. The manner of sitting as well as the time it takes to complete the task will be recorded.
Step Test | Baseline through month 12
  This is used to assess standing balance. The participant will be asked to maintain their balance on one leg while the other steps on and off a 7.5cm step as many times as possible within 15 seconds.
Walk-12 Questionnaire | Baseline through month 12
  This questionnaire is used to assess walking ability.
DM-ACTIVE Questionnaire | Baseline through month 12
  This questionnaire is used to assess the impact of DM1 on daily life.
The Physical Activity Disability Scale (PADS-R) | Baseline through month 12
  This questionnaire will assess physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Duong, PT, PhD, Principal Investigator — Stanford University; John W Day, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Universtiy, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Biogen and their collaborators will have access to coded study data. Protected Health Information (PHI)/identifiers will not be shared with Biogen or research collaborators and they will not have the key to the code linking study identification/code to the participants. When data needs to be shared, it will be via secure network using encrypted files.
Supporting Information: Study Protocol, ICF
Access Criteria: Biogen and their collaborators will have access to coded study data. PHI/identifiers will not be shared with Biogen or their collaborators, and they will not have the key linking the code to study participants.